CLINICAL TRIAL: NCT04163016
Title: A Postmarketing, Multicenter, Longitudinal, Prospective, Pharmacokinetic, Phase 1B Study in Pregnant Women With Chronic Inflammatory Diseases Treated With Cimzia (Certolizumab Pegol)
Brief Title: A Study in Pregnant Women With Chronic Inflammatory Diseases Treated With Cimzia (Certolizumab Pegol)
Acronym: CHERISH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UP0085
Record Dates: First submitted 2019-10-24; First posted 2019-11-14 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Crohn's Disease; Axial Spondyloarthritis; Plaque Psoriasis
Keywords: Cimzia; Certolizumab Pegol; Pregnant Women; Crohn's Disease (CD); Rheumatoid Arthritis (RA); Psoriatic Arthritis (PsA); Plaque Psoriasis (PSO); Axial Spondyloarthritis (AxSpA); Pharmacokinetics; CZP
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Crohn Disease; Axial Spondyloarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pharmacokinetics Sampling (Experimental): This study will include pregnant women who have decided to continue treatment with commercial certolizumab pegol (CZP) in accordance with their treating physician prior to participating in the study. Study participants will be responsible for obtaining and administering commercially available CZP under the care of their physician and according to the locally approved product label.
  From all study participants blood samples will be drawn for pharmacokinetics during the study.
  Interventions: Drug: Pharmacokinetics of certolizumab pegol

INTERVENTIONS:
Drug: Pharmacokinetics of certolizumab pegol — The collection of blood samples for pharmacokinetics (PK) is considered interventional. Blood samples will be drawn at enrollment, predose every 4 weeks (Q4W), postdose every 8 weeks (Q8W) and postpartum predose and postdose.
  Study participants will be responsible for obtaining and administering commercially available approved dosing regimens of certolizumab pegol (CZP) as prescribed by each study participant's own physician.
  Other Names: PK

SUMMARY:
The purpose of the study is to assess systemic certolizumab pegol (CZP) exposure, the formation of anti-CZP antibodies and safety of CZP across the course of pregnancy in study participants with chronic inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Participant is pregnant and ≤10 weeks gestation at the time of enrollment
* Participant must have been on stable, maintenance dose certolizumab pegol (CZP) treatment for at least 12 weeks independent of and prior to being enrolled in this study, for an approved indication in accordance with her treating physician
* Participant expects to continue CZP therapy throughout pregnancy and for at least 12 weeks postpartum
* Participant has a negative interferon gamma release assay (IGRA) or tuberculin skin test (TST) within the prior 6 months, and there has been no change in the study participant's clinical status, or social, family, or travel history. Participants with documented Bacillus Calmette-Guérin (BCG) vaccine and at low risk for tuberculosis (TB) may enroll without having a TB test performed

Exclusion Criteria:

* Participant has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Participant is not permitted to enroll into the study if she meets any of the following TB exclusion criteria:

  1. Known active TB disease
  2. History of active TB involving any organ system
  3. Latent TB infection
  4. High risk of acquiring TB infection
  5. Current nontuberculous mycobacterial (NTM) infection or history of NTM infection (unless proven to be fully recovered)
* Study participant is taking a prohibited medication or has taken a prohibited medication
* Live vaccine(s) within 1 month prior to Screening, or plans to receive such vaccines during the study
* Study participant has any clinically significant pregnancy-related clinical or test abnormality, as judged by the investigator
* Study participant had a positive or indeterminate interferon gamma release assay (IGRA) or tuberculin skin test (TST) at Screening. In case of indeterminate result, a retest is allowed if time permits; 2 results of indeterminate require exclusion of the study participant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (9):
- United States (3):
  - Up0085 104, Minneapolis, Minnesota
  - Up0085 103, Durham, North Carolina
  - Up0085 101, Oklahoma City, Oklahoma
- Up0085 500, Paris, France
- Germany (2):
  - Up0085 202, Freiburg im Breisgau
  - Up0085 201, Hamburg
- Up0085 900, Rotterdam, Netherlands
- Up0085 800, Barcelona, Spain
- Up0085 300, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in June 2020 and concluded in May 2023.
Pre-assignment Details: The Participant Flow refers to the Enrolled Set.
Groups:
- Not Dosed: This arm included participant who signed the Informed Consent Form (ICF) but withdrew from the study prior to taking a dose of commercial certolizumab pegol (CZP) after enrollment.
- CZP 200 mg Q2W: The study included pregnant women who continued treatment with commercial certolizumab pegol (CZP) in accordance with their treating physician prior to participating in the study. Study participants were responsible for obtaining and administering commercially available CZP under the care of their physician and according to the locally approved product label. Participants took commercial CZP 200 milligrams (mg) every 2 weeks (Q2W), as subcutaneous injection, during the pregnancy period (up to 40 weeks) and post-partum period (up to 13 weeks after delivery).
- CZP 400 mg Q2W: The study included pregnant women who continued treatment with commercial CZP in accordance with their treating physician prior to participating in the study. Study participants were responsible for obtaining and administering commercially available CZP under the care of their physician and according to the locally approved product label. Participants took commercial CZP 400 mg Q2W, as subcutaneous injection, during the pregnancy period (up to 40 weeks) and post-partum period (up to 13 weeks after delivery).
- CZP 400 mg Q4W: The study included pregnant women who continued treatment with commercial CZP in accordance with their treating physician prior to participating in the study. Study participants were responsible for obtaining and administering commercially available CZP under the care of their physician and according to the locally approved product label. Participants took commercial CZP 400 mg every 4 weeks (Q4W), as subcutaneous injection, during the pregnancy period (up to 40 weeks) and post-partum period (up to 13 weeks after delivery).
Period: Enrollment
Arm/Group | Not Dosed | CZP 200 mg Q2W | CZP 400 mg Q2W | CZP 400 mg Q4W
Started | 1 | 15 | 1 | 5
Completed | 0 | 15 | 1 | 5
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Treatment
Arm/Group | Not Dosed | CZP 200 mg Q2W | CZP 400 mg Q2W | CZP 400 mg Q4W
Started | 0 | 15 | 1 | 5
Completed | 0 | 12 | 1 | 3
Not Completed | 0 | 3 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Not completed — Indeterminate TB-test | 0 | 0 | 0 | 1
Not completed — Participant did not want to continue in study | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Enrolled Set (ES) which consisted of all study participants who were confirmed as having signed the Informed Consent Form (ICF) to participate in the study and had provided the first blood sample. Due to data protection/data privacy, data cannot be reported for a single participant enrolled in 'Not Dosed' and 'CZP 400 mg Q2W' arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Not Dosed | CZP 200 mg Q2W | CZP 400 mg Q2W | CZP 400 mg Q4W | Total
Number analyzed (Participants) | 0 | 15 | 0 | 5 | 20
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 0 | 15 | 0 | 5 | 20
  65 - <85 years | 0 | 0 | 0 | 0 | 0
  >=85 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 15 | 0 | 5 | 20
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 0 | 1
  White | 0 | 14 | 0 | 5 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 0 | 15 | 0 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Predose and Postdose Plasma Certolizumab Pegol (CZP) Concentrations in Women During Pregnancy, Relative to Postpartum
Description: Predose and postdose plasma CZP concentrations in women during pregnancy, relative to postpartum, were measured. The trimesters were defined as follows: Trimester 1=up to 12 weeks and 6 days gestation, trimester 2=13-28 weeks and 6 days gestation, and trimester 3=any time at or after 29 weeks gestation.
Time Frame: Predose and postdose CZP concentrations in Pregnancy trimester 1,2,3 (up to 40 weeks) and Postpartum (up to 13 weeks after delivery)
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) was a subset of the Safety Set (SS) which included those study participants for whom at least one predose or postdose sample was available which was not impacted by an important protocol deviation. Here, number analyzed signifies participants who were evaluable at specified time points. Due to data protection/data privacy, data cannot be reported for a single participant enrolled in 'CZP 400 mg Q2W' arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | CZP 200 mg Q2W | CZP 400 mg Q2W | CZP 400 mg Q4W
Number analyzed (Participants) | 15 | 0 | 4
microgram per milliliter (μg/mL)
  Predose-Trimester 1: number analyzed (Participants) | 9 | 0 | 2
  Predose-Trimester 1 | 15.251 (68.1) |  | NA (NA) — As pre-specified in the Statistical Analysis Plan, Geometric Means and Geometric Coefficient of Variation are only calculated if at least 2/3 of the concentrations are above lower limit of quantification (LLOQ) (0.032 ug/mL) and n is greater than or equal to (>=) 4. NA replaces summary statistics when the sample size is N=3 or N<3.
  Predose-Trimester 2 | 16.916 (39.9) |  | 9.027 (107.2)
  Predose-Trimester 3: number analyzed (Participants) | 11 | 0 | 4
  Predose-Trimester 3 | 16.827 (41.0) |  | 2.759 (3193.5)
  Predose-Postpartum: number analyzed (Participants) | 12 | 0 | 3
  Predose-Postpartum | 22.318 (41.1) |  | NA (NA) — As pre-specified in the Statistical Analysis Plan, Geometric Means and Geometric Coefficient of Variation are only calculated if at least 2/3 of the concentrations are above lower limit of quantification (LLOQ) (0.032 ug/mL) and n is greater than or equal to (>=) 4. NA replaces summary statistics when the sample size is N=3 or N<3.
  Postdose-Trimester 1: number analyzed (Participants) | 10 | 0 | 0
  Postdose-Trimester 1 | 20.046 (54.3) |  |
  Postdose-Trimester 2: number analyzed (Participants) | 13 | 0 | 4
  Postdose-Trimester 2 | 22.961 (44.9) |  | 46.094 (14.6)
  Postdose-Trimester 3: number analyzed (Participants) | 10 | 0 | 4
  Postdose-Trimester 3 | 25.001 (39.7) |  | 8.105 (19481.3)
  Postdose-Postpartum: number analyzed (Participants) | 12 | 0 | 3
  Postdose-Postpartum | 30.153 (47.2) |  | NA (NA) — As pre-specified in the Statistical Analysis Plan, Geometric Means and Geometric Coefficient of Variation are only calculated if at least 2/3 of the concentrations are above lower limit of quantification (LLOQ) (0.032 ug/mL) and n is greater than or equal to (>=) 4. NA replaces summary statistics when the sample size is N=3 or N<3.

2. Secondary Outcome: Number of Participants With Anti-certolizumab Pegol (CZP) Positive Antibodies Throughout the Study Period
Description: Antibodies to CZP were evaluated in plasma samples collected from all participants throughout the study. Anti-CZP antibodies (ADAb) were measured using a three-tiered assay approach: screening, confirmatory and titration assay. Samples that were confirmed as positive in the screening and confirmatory assay were evaluated in a titration assay to quantify the ADAb level and were reported as titer (reciprocal dilution factor including minimum required dilution [MRD]). Sample values that were 'positive screen' and 'positive immunodepletion' were defined as ADAb positive. Once determined positive, a study participant's highest titer was used to categorize ("titer classification") the study participant as follows: Positive less than or equal to (=)32, Positive greater than (>)32 - =128, Positive >128 - =512, Positive >512 - =1024, Positive >1024 - =4096, and Positive >4096.
Time Frame: From Enrollment to Safety Follow-up (Duration of pregnancy (up to 40 weeks) + 18 weeks) (up to 58 weeks)
Population: The Safety Set (SS) included all enrolled study participants who received at least 1 dose of CZP after Screening. Due to data protection/data privacy, data cannot be reported for a single participant enrolled in 'CZP 400 mg Q2W' arm.
Measure: Count of Participants; unit: Participants
Arm/Group | CZP 200 mg Q2W | CZP 400 mg Q2W | CZP 400 mg Q4W
Number analyzed (Participants) | 15 | 0 | 5
Participants
  Positive ≤32 | 0 |  | 0
  Positive >32 to ≤128 | 0 |  | 0
  Positive >128 to ≤512 | 1 |  | 0
  Positive >512 to ≤1024 | 0 |  | 1
  Positive >1024 to ≤4096 | 5 |  | 1
  Positive >4096 | 8 |  | 2

3. Secondary Outcome: Percentage of Participants With Adverse Events From Time of Informed Consent (Screening) Through Safety Follow-up (SFU)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical participant, temporally associated with the use of CZP, whether or not considered related to CZP.
Time Frame: From Screening to Safety Follow-up (Duration of pregnancy (up to 40 weeks) + 18 weeks) (up to 58 weeks)
Population: The SS included all enrolled study participants who received at least 1 dose of CZP after Screening. Due to data protection/data privacy, data cannot be reported for a single participant enrolled in 'Not Dosed' and 'CZP 400 mg Q2W' arms.
Measure: Number; unit: percentage of participants
Arm/Group | Not Dosed | CZP 200 mg Q2W | CZP 400 mg Q2W | CZP 400 mg Q4W
Number analyzed (Participants) | 0 | 15 | 0 | 5
percentage of participants |  | 86.7 |  | 60.0

4. Secondary Outcome: Number of Participants With Pregnancy Outcome
Description: Pregnancy outcomes were collected via a written notification by the investigator and recorded in the Pregnancy Outcome Form. Pregnancies were determined to end in delivery-live birth, delivery-still birth, spontaneous abortion, therapeutic abortion, or missing data.
Time Frame: From Enrollment to Delivery (Duration of pregnancy, up to 40 weeks)
Population: The Enrolled set included all participants who were confirmed as having signed the ICF to participate in the study and had provided the first blood sample. Due to data protection/data privacy, data cannot be reported for a single participant enrolled in 'Not Dosed' and 'CZP 400 mg Q2W' arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Not Dosed | CZP 200 mg Q2W | CZP 400 mg Q2W | CZP 400 mg Q4W
Number analyzed (Participants) | 0 | 15 | 0 | 5
Participants
  Delivery, live birth |  | 12 |  | 4
  Delivery, still birth |  | 0 |  | 0
  Spontaneous abortion |  | 0 |  | 0
  Therapeutic abortion |  | 0 |  | 0
  Missing |  | 3 |  | 1

ADVERSE EVENTS:
Time Frame: From Screening to Safety Follow-up (Duration of pregnancy (up to 40 weeks) + 18 weeks) (up to 58 weeks)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical participant, temporally associated with the use of CZP, whether or not considered related to CZP. The SS included all enrolled study participants who received at least 1 dose of CZP after Screening. Due to data protection/data privacy, data cannot be reported for a single participant enrolled in 'Not Dosed' and 'CZP 400 mg Q2W' arms.
Arm/Group | Not Dosed | CZP 200 mg Q2W | CZP 400 mg Q2W | CZP 400 mg Q4W
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/15 | 0/0 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/0 | 4/15 | 0/0 | 1/5
Other Adverse Events (participants affected / at risk) | 0/0 | 11/15 | 0/0 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Not Dosed (N=0) | CZP 200 mg Q2W (N=15) | CZP 400 mg Q2W (N=0) | CZP 400 mg Q4W (N=5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Not Dosed (N=0) | CZP 200 mg Q2W (N=15) | CZP 400 mg Q2W (N=0) | CZP 400 mg Q4W (N=5)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 6 (7) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mastitis (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perineal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Foetal vascular malperfusion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine contractions abnormal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT04163016/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT04163016/SAP_001.pdf